CLINICAL TRIAL: NCT06614153
Title: A Randomized, Open-label, Controlled, Single-dose, Multiple-dose Phase II Study to Evaluate the Pharmacokinetics,Pharmacodynamics,Efficacy and Safety of HRG2010 in Parkinson's Disease Patients With Motor Fluctuations
Brief Title: Pharmacokinetics,Pharmacodynamics,Efficacy and Safety of HRG2010 in Parkinson's Disease Patients With Motor Fluctuations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HRG2010-201
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A，Subjects will receive HRG2010(I) (Experimental): administered orally
  Interventions: Drug: HRG2010(I)
- Group B，Subjects will receive HRG2010(II) (Experimental): administered orally
  Interventions: Drug: HRG2010(II)
- Group C，Subjects will receive Sustained-release (Active Comparator): Carbidopa/Levodopa administered orally
  Interventions: Drug: Sustained-release Carbidopa/Levodopa

INTERVENTIONS:
Drug: HRG2010(I) — HRG2010(I)
  Arms: Group A，Subjects will receive HRG2010(I)
Drug: HRG2010(II) — HRG2010(II)
  Arms: Group B，Subjects will receive HRG2010(II)
Drug: Sustained-release Carbidopa/Levodopa — Sustained-release Carbidopa/Levodopa
  Arms: Group C，Subjects will receive Sustained-release

SUMMARY:
The study is a multicenter, randomized, open-label, active-controlled, Phase II clinical study. The aim of this trial is to evaluated the pharmacokinetics, pharmacodynamics,efficacy and assessed the safety of HRG2010 compared with a sustained-release cabridopa-levodopa formulation in Parkinson's Disease Patients With Motor Fluctuations.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants diagnosed at age ≥ 40 years with PD, consistent with the International Parkinson and Movement Disorder Society Clinical Diagnostic Criteria and who are being treated with stable regimens of DDCI+LD but experiencing motor fluctuations.
2. Mini Mental State Examination (MMSE) ≥ 25 at Screening Visit.
3. Hoehn and Yahr Stage II-IV when "on" at Screening Visit.
4. At Screening, the participant has predictable "Off" periods.
5. Able and willing to provide a written informed consent.

Exclusion Criteria:

1. Diagnosed with atypical or secondary parkinsonism.
2. History of narrow angle glaucoma、peptic ulcer disease or upper gastrointestinal hemorrhage.
3. Had prior functional neurosurgical treatment for PD or if such procedure(s) are planned or anticipated during the study period.
4. Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using an adequate contraceptive method.
5. In the opinion of the clinical investigator, Subjects who should not participate in the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in average percent "Off" time during waking hours at Day 33 | Last three days collected at the end of treatment period

SECONDARY OUTCOMES:
"Off" and"On" time hours during in clinic observation | Days 1 and 13
MDS-UPDRS Part III | Days 1 and 33
Change from baseline in "Off" time at Day 33 | Last three days collected at the end of treatment period
Change from baseline in the Movement Disorders Society Version of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) at Day 33 | Day 33

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided